CLINICAL TRIAL: NCT00934648
Title: An Open Label Study to Evaluate the Safety and Efficacy of Rituximab in Patients With Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Prior Treatment With Methotrexate
Brief Title: A Study of MabThera (Rituximab) in Patients With Rheumatoid Arthritis Who Have Had an Inadequate Response to Methotrexate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20546
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Results first posted 2014-06-10 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; Methotrexate

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]; Drug: methotrexate

INTERVENTIONS:
Drug: rituximab [MabThera/Rituxan] — 1000mg iv on days 1 and 15
Drug: methotrexate — 10-25mg weekly

SUMMARY:
This study will evaluate the safety and efficacy of MabThera in patients with active rheumatoid arthritis who have had an inadequate response or were intolerant to treatment with methotrexate. Eligible patients will receive MabThera (1000mg by intravenous infusion) on days 1 and 15, and background methotrexate (oral or subcutaneous dose of 10-25mg weekly). After the initial study period of 24 weeks, eligible patients may receive up to 3 re-treatments with MabThera. The anticipated time on study treatment is 1-2 years, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* receiving out-patient treatment;
* experienced an inadequate response to previous or current treatment with methotrexate.

Exclusion Criteria:

* rheumatic autoimmune disease other than RA, or significant systemic involvement secondary to RA;
* history of, or current, inflammatory joint disease other than RA;
* previous treatment with any cell-depleting therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Morocco (4):
  - Casablanca
  - Marrakesh
  - Rabat
  - Salé

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab 1000 Milligrams (mg): Participants received rituximab 1000 mg administered intravenously (IV) and methylprednisolone 100 mg, IV, on Days 1 and 15; all participants were receiving background methotrexate (MTX) 10-25 mg weekly by mouth or parenterally per local prescribing guidelines.
Period: Overall Study
Arm/Group | Rituximab 1000 Milligrams (mg)
Started | 15
Completed | 6
Not Completed | 9
Not completed — Failure to return | 8
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population: all participants who received any part of an infusion.
Groups:
- Rituximab 1000 mg: Participants received rituximab 1000 mg administered IV and methylprednisolone 100 mg, IV, on Days 1 and 15; all participants were receiving background MTX 10-25 mg weekly by mouth or parenterally per local prescribing guidelines.
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Adverse Event (AE)
Time Frame: Week 104
Population: Safety population: included all participants who have received any part of an infusion of the study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 15
percentage of participants | 26.7

2. Secondary Outcome: Disease Activity Score Based on 28-Joint Count (DAS28)
Description: DAS28 was calculated from the number of swollen joints and tender joints using the 28 joint count; the erythrocyte sedimentation rate (ESR) measured in millimeters per hour [mm/hr]); and the Patient's Global Assessment of disease activity (participant-rated visual analog assessment [VAS]) with transformed scores with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity. Overall, a DAS28 score of less than or equal to (≤) 3.2 equals (=) low disease activity, and a DAS28 score of greater than (>) 3.2 to 5.1 = moderate to high disease activity.
Time Frame: Day 1 and Week 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 15
scores on a scale
  Day 1 | 5.79 (1.03)
  Week 24 | 4.41 (1.88)

3. Secondary Outcome: Percentage of Participants With a DAS28 Response by European League Against Rheumatism (EULAR) Category
Description: DAS28-based EULAR response criteria were used to measure individual response as no response, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline greater than (>)1.2 with DAS28 less than or equal to (≤)3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to ≤5.1 or change from baseline >0.6 to ≤1.2 with DAS28 ≤5.1; non-responders: change from baseline ≤0.6 or change from baseline >0.6 and ≤1.2 with DAS28 >5.1.
Time Frame: Screening, Day 1, and Weeks 24 and 104
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 15
percentage of participants
  ≤3.2 at Screening | 0
  >3.2 and ≤5.1 at Screening | 22.2
  >5.1 at Screening | 77.8
  ≤3.2 at Day 1 | 0
  >3.2 and ≤5.1 at Day 1 | 33.3
  >5.1 at Day 1 | 66.7
  ≤3.2 at Week 24 | 37.5
  >3.2 and ≤5.1 at Week 24 | 37.5
  >5.1 at Week 24 | 25.0
  ≤3.2 at Week 104 | 33.3
  >3.2 and ≤5.1 at Week 104 | 33.3
  >5.1 at Week 104 | 33.3

4. Secondary Outcome: Percentage of Participants With Changes in Bone Density
Description: Change in bone density in participants untreated with bisphosphonates was classified as percentage of participants with osteoporosis, osteopenia, or normal. In some participants, no determinations were available.
Time Frame: Screening, Weeks 48 and 104
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 15
percentage of participants
  Osteoporosis, Screening | 20
  Osteopenia, Screening | 46.7
  Normal, Screening | 0
  Not determined, Screening | 33.3
  Osteoporosis, Week 48 | 6.7
  Osteopenia, Week 48 | 13.3
  Normal, Week 48 | 6.7
  Not determined, Week 48 | 73.3
  Osteoporosis, Week 104 | 0
  Osteopenia, Week 104 | 40
  Normal, Week 104 | 0
  Not determined, Week 104 | 60

ADVERSE EVENTS:
Time Frame: Adverse events were collected from signing of informed consent through the end of the follow-up period (Week 104).
Arm/Group | Rituximab 1000 mg
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 4/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab 1000 mg (N=15)
Fever (General disorders) | 1
Scalp infection (Infections and infestations) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash of face (Skin and subcutaneous tissue disorders) | 1
Diffuse skin rash (Skin and subcutaneous tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Tightening of throat and tongue (Respiratory, thoracic and mediastinal disorders) | 1
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.